CLINICAL TRIAL: NCT02650999
Title: Phase I/II Study of Pembrolizumab in Patients Failing to Respond to or Relapsing After Anti-CD19 Chimeric Antigen Receptor Modified T Cell Therapy for Relapsed or Refractory CD19+ Lymphomas
Brief Title: Pembrolizumab in Patients Failing to Respond to or Relapsing After CAR T Cell Therapy for Relapsed or Refractory Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 46415
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: CD19+ Diffuse Large B-cell Lymphomas; Follicular Lymphomas; Mantle Cell Lymphomas
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Single arm, pembrolizumab 200mg IV every 3 weeks until progression/toxicity
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg intravenously (IV)

SUMMARY:
Single center, phase I/II trial of pembrolizumab after CTL019 for CD19+ lymphomas. Patients will have CD19+ diffuse large B-cell, follicular, or mantle cell lymphomas relapsed/refractory after CTL019. 12 total patients will be enrolled. Safety of pembrolizumab (primary endpoint) will be determined using a Bayesian monitoring rule for treatment-related adverse events causing drug discontinuation. Secondary efficacy endpoints include overall response rate and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma grade 1-3A, diffuse large B cell lymphoma, and mantle cell lymphoma by World Health Organization 2009 classification
* Relapsed/refractory lymphoma after CTL019 - Be willing and able to provide written informed consent/assent for the trial.
* Age 18 years or older on day of signing informed consent.
* Have baseline imaging within 6 weeks of enrollment (CT, MR or PET/CT imaging) and have measurable disease on physical examination or imaging studies.

  -- Not pregnant or breastfeeding
* Any lesion 1.5 cm in long axis dimension is considered measurable.
* Performance status of 0-2 on the ECOG Performance Scale
* Demonstrate adequate organ function.
* Absolute neutrophil count (ANC) ≥1,000 /mcL
* Platelets≥50,000 / mcL
* Hemoglobin ≥8 g/dL without transfusion or EPO dependency (within 7 days of assessment)
* Serum creatinine OR Measured or calculated a creatinine clearance (aCreatinine clearance should be estimated per institutional standard) (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment. An exception will be made for patients who have received CTL019/CTL119 on experimental protocol; these patients will be eligible to enroll once progression of disease or failure to respond is documented by clinical or radiologic assessment.
2. Patient has received intervening therapy for lymphoma after CTL019/CTL119 infusion.
3. Has active cytokine release syndrome from CTL019/CTL119 infusion.
4. Has a known history of active TB (Bacillus Tuberculosis).
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Toxicities that are disease related will not exclude patients.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention in the opinion of the Principal Investigator prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Has a history of (non-infectious pneumonitis that required steroids or has current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02-25 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Schuster, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chong EA, Alanio C, Svoboda J, Nasta SD, Landsburg DJ, Lacey SF, Ruella M, Bhattacharyya S, Wherry EJ, Schuster SJ. Pembrolizumab for B-cell lymphomas relapsing after or refractory to CD19-directed CAR T-cell therapy. Blood. 2022 Feb 17;139(7):1026-1038. doi: 10.1182/blood.2021012634. PMID 34496014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Pembrolizumab: 200mg intravenously (IV)
Arm/Group | Single Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Percentage of subjects who discontinued therapy due to dose-limiting toxicity
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Single Arm
Number analyzed (Participants) | 12
percentage of subjects | 8.33 [0.4 to 40.2]

2. Secondary Outcome: Overall Response Rates
Description: 3 months Overall response rates
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Single Arm
Number analyzed (Participants) | 12
percentage of subjects | 25 [6.7 to 57.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 2.5 years, from the initiation of the first patient on therapy (June 7, 2016) through treatment of the last patient (January 11, 2019). All adverse events on individual patients were recorded from the time of first dose of pembrolizumab through completion of the Safety Follow Up Visit. SAEs that occured within 90 days of the end of treatment or before initiation of a new anti-cancer treatment were also followed and recorded.
Description: Adverse events were collected by trained research nurse, with attributions assigned by Investigating physician. AEs were recorded in cumulative AE tables, with final review by Principal Investigator at the conclusion of each subject's trial participation.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=12)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
acidosis (Metabolism and nutrition disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cytokine Release Syndrome (Immune system disorders) | 1
blood bilirubin increased (Hepatobiliary disorders) | 1
sepsis (Infections and infestations) | 1
hypercalcemia (Investigations) | 1
delirium (Psychiatric disorders) | 1
fever (General disorders) | 1
other: odynophagia (Gastrointestinal disorders) | 1 — odynophagia
dysphagia (Gastrointestinal disorders) | 1
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
optic disorder (Eye disorders) | 1
non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=12)
tachycardia (Cardiac disorders) | 1
atrial fibrillation/atrial flutter (Cardiac disorders) | 1
nausea (Gastrointestinal disorders) | 5
diarrhea (Gastrointestinal disorders) | 3
vomiting (Gastrointestinal disorders) | 3
dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
GI disorders, other: odynophagia (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
fatigue (General disorders) | 6
fever (General disorders) | 4
infusion related reaction (General disorders) | 1
lower extremity edema (General disorders) | 1
Facial pain (General disorders) | 1
Facial edema (left side) (General disorders) | 1
Flank pain (General disorders) | 1
Flu-like symptoms (General disorders) | 1
gait disturbance (General disorders) | 1
Infections, other: Zoster (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
urinary tract infection (Infections and infestations) | 1
Neutropenia (Investigations) | 4
Lymphocyte count decreased (Investigations) | 7
Anemia (Investigations) | 4
INR increased (Investigations) | 2
AST elevated (Investigations) | 5
ALT elevated (Investigations) | 4
thrombocytopenia (Investigations) | 2
alkaline phosphatase elevated (Investigations) | 1
PTT prolonged (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
WBC decreased (Investigations) | 3
Investigations - Other, Platelets elevated (Investigations) | 1
Investigations - Other, WBC increased (Investigations) | 1
Investigations - Other, ANC increased (Investigations) | 1
Weight loss (Investigations) | 1
Investigations, other: low serum total protein (Investigations) | 1
Investigations, other: elevated urine pH (Investigations) | 1
Investigations, other: elevated MHC (Investigations) | 1
Investigations, other: elevated CO2 (Investigations) | 1
Blood LDH increased (Investigations) | 1
hyperglycemia (Metabolism and nutrition disorders) | 4
hypoglycemia (Metabolism and nutrition disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 3
hypokalemia (Metabolism and nutrition disorders) | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 2
hypophosphatemia (Metabolism and nutrition disorders) | 3
hypocalcemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
dehydration (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - other, phosphorus elevated (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Synovitis (MCP, middle finger, left hand) (Musculoskeletal and connective tissue disorders) | 1
pain (back, buttock, right leg / sciatica distribution) (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3
Lower back pain (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Post-herpetic neuralgia (Nervous system disorders) | 1
Nervous system - Other, cauda equina syndrome (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
urinary hesitancy (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
urinary retention (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 3
Skin disorders, other: inflammation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT02650999/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT02650999/ICF_001.pdf